CLINICAL TRIAL: NCT00074724
Title: Dobutamine Echocardiography In Patients With Ischemic Heart Failure Evaluated for Revascularization
Acronym: DECIPHER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 153; 1R01HL070011-01A1 (NIH)
Record Dates: First submitted 2003-12-19; First posted 2003-12-23 (Estimated); Results first posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2016-06

CONDITIONS: Cardiovascular Diseases; Coronary Disease; Heart Failure; Heart Failure, Congestive; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Disease; Heart Failure; Heart Diseases | interventions — Coronary Artery Bypass; Echocardiography, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Medical Therapy (Active Comparator): All medical interventions know to improve outcomes in patients with ischemic left ventricular dysfunction.
  Interventions: Drug: Modern medical management; Device: Dobutamine echocardiography; Drug: Optimal medical therapy
- CABG (Active Comparator): Surgical revascularization in conjunction with optimal medical therapy.
  Interventions: Procedure: Coronary Artery Bypass; Device: Dobutamine echocardiography

INTERVENTIONS:
Procedure: Coronary Artery Bypass — coronary revascularization using arterial or vein conduits
  Other Names: CABG
  Arms: CABG
Drug: Modern medical management — Therapies with evidence-based recommendations.
  Other Names: Optimal medical therapy
  Arms: Medical Therapy
Device: Dobutamine echocardiography — Incremental dose administration of dobutamine to elicit a contractile response of the myocardium.
  Other Names: dobutamine echo
Drug: Optimal medical therapy — All medical interventions known to improve outcomes in patients with ischemic left ventricular dysfunction.
  Other Names: MOdern medical therapy
  Arms: Medical Therapy

SUMMARY:
To define the role of the assessment of myocardial viability with dobutamine echocardiography (DE) in the clinical evaluation and selection of the best treatment for a high-risk subset of patients with coronary artery disease.

DETAILED DESCRIPTION:
BACKGROUND:

The number of individuals presenting with coronary artery disease (CAD) with impaired left ventricular (LV) function (measured as ejection fraction {EF}<35%), and clinical evidence of heart failure (HF) continues to increase. Patients with these conditions face the need for continuous and intensive medical management and poor quality of life. The STICH trial is designed to compare medical management to surgical revascularization in these patients. STICH's design includes myocardial function determination by several methods. The timely and important question of myocardial viability when function is poor is being examined using radionuclide methods. However, there is no consensus on the best technique to determine myocardial viability, or data to support this assessment as a potential determinant of prognosis following surgery. DECIPHER STICH adds dobutamine echocardiography (DE) for myocardial viability measurement to the parent trial. The study is of significance by addressing an important question and adding data for a technique that bears approximately half the cost of radionuclide methods. Furthermore, the revised design will allow for randomized and blinded evaluations of different treatment modalities according to myocardial viability determined by two different techniques.

DESIGN NARRATIVE:

The Dobutamine Echocardiography in Patients with Ischemic Heart failure Evaluated for Revascularization Study, as part of the Surgical Treatment for Ischemic Heart Failure Trial (DECIPHER-STICH), is designed to address the hypothesis that assessment of myocardial viability with dobutamine echocardiography (DE) in patients with coronary artery disease (CAD), left ventricular (LV) dysfunction and heart failure (HF) identifies the patients who derive the greatest survival benefit from surgical revascularization over medical therapy. In addition, this study will determine the value of DE for the prediction of recovery of LV function following revascularization, the clinical value of DE relative to that of radionuclide techniques used for the same purpose, and the relationship between abnormal LV size and shape and the contractile reserve of dysfunctional myocardium.

DECIPHER-STICH is an ancillary study to the large-scale STICH trial, a multicenter international randomized study designed to define the role of coronary artery bypass grafting (CABG) and surgical ventricular restoration (SVR) in the treatment of HF in patients with CAD and LV dysfunction. In previous studies, DE has compared favorably to other methods for the detection of viable myocardium. The widespread availability of echocardiography and the possibility of simultaneously deriving information about structural abnormalities (e.g., thrombi), valve function, and intracardiac pressures in addition to the real-time assessment of regional and global systolic function make DE particularly useful for the comprehensive evaluation of CAD patients with LV dysfunction. Because patients in the STICH trial will also undergo radionuclide tests, the DECIPHER-STICH study will allow a comparison of the most commonly used techniques for assessment of myocardial viability. Patients recruited into the STICH trial will be invited to participate in the DECIPHER-STICH study and asked to sign a separate consent form prior to the randomized assignment of therapy. Forty centers from North America and Europe recruiting patients into the STICH trial have agreed to take part in the DECIPHER-STICH study. A total of 1,450 of the 2,800 patients enrolled into the STICH trial will undergo DE prior to treatment. DECIPHER-STICH will address the hypothesis of greater beneficial effect of coronary artery bypass surgery (CABG) over medical therapy alone on 3-year survival rate with 80% power to detect a 25%-to-12.5% reduction in all-cause mortality in patients with viable myocardium. In addition, the study will have >99% power to address three important secondary hypotheses. The results of this study will provide definitive information regarding the value of assessing myocardial viability with DE and significant clinical implications for the selection of patients with CAD, LV dysfunction, and HF who are most likely to benefit from surgical revascularization.

ELIGIBILITY:
Enrollment Requirements

Inclusion Criteria:

* Symptomatic heart failure defined as NYHA Class II - IV (within 3 months of entry)
* LV less than 35% defined by CMR or gated SPECT studies
* Coronary anatomy suitable for revascularization

Exclusion Criteria:

* Primary valvular heart disease clearly defined indicating the need for valve repair or replacement
* Patients with concurrent cardiogenic shock or requiring inotropic or intra-aortic balloon support
* PCI planned for CAD treatment
* Acute myocardial infarction within 30 days
* More than one prior cardiac operation
* Non-cardiac illness with life expectancy of less than 3 years
* Non-cardiac illness imposing substantial operative mortality. Patients eligible to enter the study will be further evaluated by the STICH team for SVR eligibility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2003-05 (Actual); Primary Completion 2008-12 (Actual); Study Completion 2017-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julio Panza, Principal Investigator — Medstar Health Research Institute

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Medical Therapy | CABG
Started | 0 (The PI has left the institution and no results data is available. Efforts were made to contact the PI/study team members, as well as to review data on shared drives, IRB historical records and published resources, but were unsuccessful. No study data are available) | 0 (The PI has left the institution and no results data is available. Efforts were made to contact the PI/study team members, as well as to review data on shared drives, IRB historical records and published resources, but were unsuccessful. No study data are available)
Completed | 0 (The PI has left the institution and no results data is available. Efforts were made to contact the PI/study team members, as well as to review data on shared drives, IRB historical records and published resources, but were unsuccessful. No study data are available) | 0 (The PI has left the institution and no results data is available. Efforts were made to contact the PI/study team members, as well as to review data on shared drives, IRB historical records and published resources, but were unsuccessful. No study data are available)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The PI has left the institution and no results data is available. Efforts were made to contact the PI/study team members, as well as to review data on shared drives, IRB historical records and published resources, but were unsuccessful. No study data are available
Groups:
- Total: Total of all reporting groups
Arm/Group | Medical Therapy | CABG | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Age, Continuous
Sex: Female, Male

OUTCOME MEASURES:

1. Primary Outcome: Survival Free of Cardiac Hospitalization
Time Frame: 3 years
Population: as for baseline characteristics
Arm/Group | Medical Therapy | CABG
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Left Ventricular Ejection Fraction
Time Frame: 4 months and 2 years
Population: as for baseline characteristics
Arm/Group | Medical Therapy | CABG
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: The PI has left the institution and no results data is available. Efforts were made to contact the PI/study team members, as well as to review data on shared drives, IRB historical records and published resources, but were unsuccessful. No study data are available
Description: The PI has left the institution and no results data is available. Efforts were made to contact the PI/study team members, as well as to review data on shared drives, IRB historical records and published resources, but were unsuccessful. No study data are available
Arm/Group | Medical Therapy | CABG
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No